CLINICAL TRIAL: NCT06964100
Title: Exploring the Relationship Between Heart Rate Variability (HRV), Training Load, and Endurance Performance
Status: Recruiting | Type: Observational
Sponsor: PepsiCo Global R&D (Industry)
Responsible Party: Sponsor
Other Study IDs: PEP-2502
Record Dates: First submitted 2025-04-15; First posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-04

CONDITIONS: Heart Rate Variability
Keywords: heart rate variability; HRV; real world; activity tracker; app engagement; app functionality; remote

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The ability of smart phones, aided by wearable devices (e.g. smart watches), to collect a variety of data, including physical activity, heart rate, and other exercise metrics, may provide a unique opportunity to understand real-world variability. The primary objective of this study is to test user engagement, app functionality, and feasibility of the newly developed Gatorade Sports Science Institute (GSSI) Labs App to conduct Real-World research studies. The secondary purpose of this study is to determine if Training Intensity (%Heart Rate maximum) in minutes during low heart rate variability (HRV) periods (below HRV baseline consecutive days) will have a negative relationship with post-study 5K (5 kilometer) running times as measured by their activity tracker, which could lead to personalized training recommendations using HRV. This study is conducted remotely, there are no in-person visits.

DETAILED DESCRIPTION:
Heart rate variability (HRV) is an indirect biomarker of an individual's performance readiness and recovery. HRV is a ubiquitous biomarker measured by most consumer-grade wearable fitness trackers. However, there is little documented on the relationship between HRV, training load, and performance measures in the Real-World. Using activity trackers to monitor multiple physiological and subjective measures of health and wellness, subjects will perform self-administered 5 kilometer (5K) timed runs on Week 1, Week 4, and Week 8. Users will be instructed to run their 5K (3.1 miles) on the same outdoor course, indoor track, or treadmill to provide consistency in their performance assessments, with the understanding that there will be some limitations in creating a consistent performance assessment environment (i.e.; weather).

ELIGIBILITY:
Inclusion Criteria:

Actively participating in cardiovascular training (3-5 days/week).

Able to run a 5K (3.1 miles) distance at a self-selected location, three times over 8 weeks.

Age 18-65 years.

Subject is willing to refrain from vigorous exercise (light physical activity only) 24 hours prior to timed 5K assessment.

Subject is willing to avoid alcohol consumption 24 hours prior to 5K assessment.

Subject is willing to provide consent.

Subject is able to continuously wear their activity tracker, including during sleep, except when submerged underwater (i.e., swimming, bathing).

Subjects must have compatible wearable device (Android, Apple Health, Dexcom, Fitbit, Garmin, Health Connect, Oura, Polar, Whoop, and Withings).

Exclusion Criteria:

Individual has a condition the Investigator believes would interfere with his ability to provide informed consent, comply with the project/study protocol, which might confound the interpretation of the project/study results or put the person at undue risk.

Those with a medical history that would interfere with the results of this study.

Those that have ≥1 risk factor for cardiovascular disease according to the American College of Sports Medicine.

Age: Men ≥ 45 yrs; Women ≥ 55 yrs.

Family History: Heart attack, "bypass surgery", or sudden death before the age of 55 yrs for father/brother, or before 65 yrs for mother/sister.

Cigarette Smoking: Current smoker, or have quit < 6 months, or exposed to environmental smoke.

Sedentary lifestyle: Not participating in moderate (sweating) physical activity at least 3 days/week for 3-months.

Obesity: Body mass index ≥ 30 kg/m2 or waist girth 102 cm (40 inches) for men and 88 cm (35 inches) for women.

Hypertension: Systolic Blood Pressure ≥ 140 mmHg and/or Diastolic ≥90 mmHg, or taking medication.

Dyslipidemia: LDL ≥130 mg/dl, or HDL < 40 mg/dl, or taking medication. Or triglycerides (TG) > 200 > mg/dl.

Pre-diabetes: Impaired fasting glucose (IFG) ≥ 100 mg/dl or oral glucose tolerance test (OGTT) ≥ 140 or ≤ 199 mg/dl confirmed by two different measurements.

Under the care of a physician.

Sleep disorders.

Using prescription medications that would impact sleep.

If female, you are not pregnant, planning to get pregnant or currently breast feeding.

Not able to wear activity tracker continuously.

Lack of proficiency in English.

Lack of proficiency or access to the internet and email address.

Participation in another clinical trial within the past 30 days.

Subject is employed by, or has a parent, guardian, or other immediate family member employed by a company that manufactures any products that compete with any Gatorade product. If subject is unsure if a company would be considered a competitor to Gatorade, they will be asked to please let the study investigator know the name of the other company and the nature of their relationship to that company before they sign the informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers ages 8-65, actively participating in cardiovascular training (3-5 days/week), able to run a 5K (3.1 miles) distance at a self-selected location, three times over 8 weeks, wear an activity tracker and willing to use the study smartphone app.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-04-04 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
User engagement with Gatorade Sports Science Institute (GSSI) Labs app | From activating app through study Week 8
  Percent (%) who complete enrollment, informed consent form (ICF), demographics, sync biometrics, complete journal entries, 5 kilometer (5K) performance assessment, and complete study

SECONDARY OUTCOMES:
Pre-, Mid-, and Post-5K run times and wearable activity tracker biometrics: Heart rate variability (HRV) | Week 1 baseline, Week 4 and Week 8
  Fluctuation in the amount of time between heartbeats in milliseconds (ms)
Pre-, Mid-, and Post-5K run times and wearable activity tracker biometrics: Resting heart rate (RHR) | Week 1 baseline, Week 4 and Week 8
  Heart rate at rest in beats per minute (bpm)
Pre-, Mid-, and Post-5K run times and wearable activity tracker biometrics: Sleep Quantity | Week 1 baseline, Week 4 and Week 8
  Sleep at night in minutes
Pre-, Mid-, and Post-5K run times and wearable activity tracker biometrics: Sleep Efficiency | Week 1 baseline, Week 4 and Week 8
  Percentage (%) of time spent asleep while in bed, calculated by dividing total sleep time by time in bed in hours
Pre-, Mid-, and Post-5K run times and wearable activity tracker biometrics: Sleep Consistency | Week 1 baseline, Week 4 and Week 8
  Percent (%) of consistency in sleep-wake schedule
Pre-, Mid-, and Post-5K run times and wearable activity tracker biometrics: Training Zones Percent (%) maximum heart rate (HRmax) in minutes | Week 1 baseline, Week 4 and Week 8
  Heart rate training zones from Zone 1 (Very Light/Recovery): 50-60 percent (%) of maximum heart rate (HR) to Zone 5 (Very Hard/Maximum): 90-100% of max HR, in minutes (min)

OTHER OUTCOMES:
Estimated VO2 Max | At baseline
  Maximal oxygen consumption (VO2 max) = 15.3 x (HRmax/HRrest)
Demographics | At enrollment
  Age, Gender, Race
Activity details | During study period from Baseline Week 1 to Week 8
  Journal entries (Felt nervous or anxious, Have any alcoholic drinks, Have caffeine, Feel emotionally and mentally stable, Feel energized, Hydrated sufficiently, Take melatonin, Feel motivated, Felt recovered, Feeling sick or ill, and Feel stress).

CONTACTS AND LOCATIONS:
Overall Officials: Corey Ungaro, do not contact to enroll, PhD, Principal Investigator — PepsiCo R&D Life Sciences, Sports Science
Locations (1):
- Remote study, no physical site. Managed by Gatorade Sports Science Institute. Do not contact investigators to enroll. Recruitment is handled by an independent agency., Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No